CLINICAL TRIAL: NCT06088810
Title: The Impact of Music Intervention on Sleep: CoMPoSER Trial
Brief Title: The Impact of Music Intervention on Sleep
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PRO00115115; 1K23AG073618-01 (NIH)
Record Dates: First submitted 2023-09-26; First posted 2023-10-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Dementia
Keywords: Dementia
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The study will consist of 144 participants (72 dyads). Dyads will receive 4 weekly phone calls in addition to the baseline and post-intervention in-person home visits. Those receiving the CoMPoSER intervention will undergo the following components: A) relaxation techniques; B) meaningful and relaxing music playlist, tailored to PLWD preferred genre, and C) nighttime routine guidance. Those undergoing the attention control intervention will receive sleep education. The attention control design includes participants finding their own treatment if assigned to no-treatment group and higher study dropout rates.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Education Group (Active Comparator): Participants in this group will receive sleep education.
  Interventions: Other: Sleep Education
- CoMPoSER Intervention Group (Experimental): Participants in this group will use a mobile application that plays calming music personalized for sleep enhancement.
  Interventions: Other: CoMPoSER intervention group

INTERVENTIONS:
Other: CoMPoSER intervention group — Participants in the intervention will use a mobile application that plays calming music personalized for sleep enhancement, relaxation techniques and nighttime routine guidance.
  Arms: CoMPoSER Intervention Group
Other: Sleep Education — Participants in this intervention will receive sleep education based on the NIH/NIA guide, which includes tips for getting a good night's sleep.
  Arms: Sleep Education Group

SUMMARY:
The primary purpose of this Stage 1b NIH-funded clinical trial (K23AG073618, PI Petrovsky) is to determine the efficacy of a 1-month music intervention (Calming Music Personalized for Sleep Enhancement in PeRsons living with Dementia, CoMPoSER) on health outcomes in 72 dyads (144 participants) of persons living with dementia (PLWD) and their caregivers (Stage 1b). The secondary purpose of this research project is to examine the mechanism of stress reduction and sustained effects of the music intervention on PLWD and caregiver well-being. We will evaluate the acceptability of the mobile application CoMPoSER in a pilot RCT and determine the impact of the mobile application CoMPoSER on PLWD (sleep latency, sleep efficiency, wake after sleep onset, total sleep time, sleep quality) and caregiver (perceived stress and well-being) outcomes.

DETAILED DESCRIPTION:
Aim 1: Evaluate the acceptability of the mobile application CoMPoSER in a pilot RCT.

Aim 2: Determine the impact of the mobile application CoMPoSER on PLWD (sleep latency, sleep efficiency, wake after sleep onset, total sleep time, sleep quality) and caregiver (perceived stress and well-being) outcomes.

Aim 3: Examine stress reduction as a mechanism of action measured via salivary cortisol by which 1-month long CoMPoSER intervention affects insomnia symptoms in PLWD.

Aim 4: To determine the sustained (3 months) efficacy of CoMPoSER compared to control group on PLWD and caregiver health outcomes.

ELIGIBILITY:
Inclusion Criteria for persons living with dementia (PLWD):

* Age 60 and above
* Existing physician diagnosis of dementia or self-reported memory impairment and Clinical Dementia Rating Scale score of greater than 0.5,
* Score of >10 on the Insomnia Severity Index
* Stable dose of psychotropic medications
* Agreeing to wear an actiwatch for the duration of the study

PLWD Exclusion Criteria:

* Hearing impairment
* Planned transition to a residential or institutional care facility in 3 months
* Presence of extrapyramidal symptoms or acute sleep disruption
* Bed bound
* Living in an alternative home setting (such as Assisted Living Community)

Informal caregivers inclusion criteria:

* Age 18 and above.
* Providing at least 4 hours of daily care
* Living with PLWD
* Able to read and communicate in English

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | 4 weeks
  At least 80% of the dyads will find the intervention acceptable

SECONDARY OUTCOMES:
PLWD Objective Sleep Outcomes | 1 month, 3 months
  Compared to PLWD in the sleep education control group, PLWD in the CoMPoSER intervention will experience improved insomnia symptoms of sleep latency, sleep efficiency, wake after sleep onset, total sleep time measured via sleep diary and actigraphy.
PLWD Subjective Sleep Outcomes | 1 month, 3 months
  Compared to PLWD in the sleep education control group, PLWD in the CoMPoSER intervention will experience improved sleep quality via self-report. The Pittsburgh Sleep Quality Index (PSQI) will be used to measure sleep quality. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty). The component scores are summed to produce a global score (range 0 to 21). Higher scores indicate worse sleep quality.
Caregiver Stress Outcome | 1 month, 3 months
  Compared to caregivers in the sleep education control group, caregivers in the CoMPoSER intervention will experience less perceived stress. The Perceived Stress Scale (PSS) will be used to assess perceived stress among caregivers. The PSS has 10 items. Individual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
Caregiver Wellbeing Outcome (Burden) | 1 month, 3 months
  Compared to caregivers in the sleep education control group, caregivers in the CoMPoSER intervention will experience improved wellbeing (less burden). The Zarit Burden Scale will be used to assess caregiver wellbeing. The ZBI consists of 22 items rated on a 5-point Likert scale that ranges from 0 (never) to 4 (nearly always) with the sum of scores ranging between 0-88. Higher scores indicate greater burden/worse wellbeing.
Caregiver Wellbeing Outcome (Depression) | 1 month, 3 months
  Compared to caregivers in the sleep education control group, caregivers in the CoMPoSER intervention will experience improved wellbeing (less depression). The Patient Health Questionnaire (PHQ-9) will be used to assess caregiver wellbeing (depression). The PHQ-9 consists of 9 items rated on a 4-point Likert scale that ranges from 0 (not at all) to 4 (nearly every day) with the sum of scores ranging between 0-27. Higher scores indicate greater depression/worse wellbeing.
Stress Change | 1 month
  Changes in diurnal salivary cortisol from baseline to 1 month will mediate the effect of CoMPoSER on insomnia symptoms in PLWD.

CONTACTS AND LOCATIONS:
Overall Officials: Darina Petrovsky, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vitiello MV, Borson S. Sleep disturbances in patients with Alzheimer's disease: epidemiology, pathophysiology and treatment. CNS Drugs. 2001;15(10):777-96. doi: 10.2165/00023210-200115100-00004. PMID 11602004
- [Background] Petrovsky DV, Ramesh P, McPhillips MV, Hodgson NA. Effects of music interventions on sleep in older adults: A systematic review. Geriatr Nurs. 2021 Jul-Aug;42(4):869-879. doi: 10.1016/j.gerinurse.2021.04.014. Epub 2021 Jun 2. PMID 34090233
- [Background] Cheour S, Cheour C, Kilani C, Guemri A, Zineddine D, Khelifa R, Supriya R, Bragazzi NL, Cheour F, Baker JS, Gaied-Chortane S. Salivary Testosterone and Cortisol Levels in Tunisian Elderly Male Patients With Mild Alzheimer's Disease. Implications of Musical Therapy And/Or Physical Rehabilitation. Front Physiol. 2022 Aug 5;13:839099. doi: 10.3389/fphys.2022.839099. eCollection 2022. PMID 35991172
- [Background] Takahashi T, Matsushita H. Long-term effects of music therapy on elderly with moderate/severe dementia. J Music Ther. 2006 Winter;43(4):317-33. doi: 10.1093/jmt/43.4.317. PMID 17348758
- [Background] Gooneratne NS, Vitiello MV. Sleep in older adults: normative changes, sleep disorders, and treatment options. Clin Geriatr Med. 2014 Aug;30(3):591-627. doi: 10.1016/j.cger.2014.04.007. Epub 2014 Jun 12. PMID 25037297
- [Background] Shum A, Taylor BJ, Thayala J, Chan MF. The effects of sedative music on sleep quality of older community-dwelling adults in Singapore. Complement Ther Med. 2014 Feb;22(1):49-56. doi: 10.1016/j.ctim.2013.11.003. Epub 2013 Nov 14. PMID 24559816